CLINICAL TRIAL: NCT06414928
Title: In-hospital & 30-day Prognostication of Acute Heart Failure Patients by Comparing 4 Validated Scores in Patients Presenting to the Emergency Department of Cardiac Tertiary Care Hospital, Karachi- Pakistan
Brief Title: Prognostic Model Heart Failure
Status: Recruiting | Type: Observational
Sponsor: National Institute of Cardiovascular Diseases, Pakistan (Other)
Responsible Party: Principal Investigator, Madiha Fatima, Senior Registrar Emergency, National Institute of Cardiovascular Diseases, Pakistan
Other Study IDs: IRB-63/2023
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Acute Heart Failure — Consecutive patients presented at Emergency Departement with Acute Heart Failure

SUMMARY:
This study aims to determine the prognosis of heart failure in our population by using multiple validated risk scores and to evaluate the strengths of these scores in assessing prognosis with better discrimination.

DETAILED DESCRIPTION:
After fulfilling the eligibility criteria, informed consent will be obtained from all the patients regarding using data for research while maintaining anonymity. All the included patients will be interviewed by the assigned physician to complete the detailed questionnaire, including patient demographics, risk factors, and validated questionnaires including the Acute Decompensated Heart Failure National Registry (ADHERE), The Get With The Guideline-Heart Failure (GWTG-HF) Risk Score, the Ottawa Heart Failure Risk Scale (OHFRS), and EHMRG30-ST score. All the patients will be followed after 30 days, and survival status will be obtained. The AUC of the GWTG-HF risk score for all-cause death was 0.687 (95% CI, 0.649-0.725) [18], at 95% confidence interval, ±3% margin of error, the sample size was calculated to be n=626 patients. The calculated sample size was inflated by a factor of 1.5 for the design effect; hence, the sample size for the study will be N=939.

For data verification, 10% of the data will be cross-checked with the source document (Patient file).

ELIGIBILITY:
Inclusion Criteria:

* Patients of age > 18 years or more
* Either gender
* Patients visited the emergency department at NICVD, Karachi
* Newly/Already diagnosed with Heart Failure
* Giving informed consent
* Who can be followed in 30 days via Telephone or in OPD

Exclusion Criteria:

* Patients of age <18 years
* Patients who do not give consent
* Patients who are mentally handicapped due to any neurological or psychiatric illness (excluding depression/anxiety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presented at the Emergency Department with signs and symptoms of Acute Heart Failure who are fulfilling the eligibility criteria will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
In-Hospital Prognosis | From admission till discharge/death
  Factors affecting in-hospital prognosis of patients with acute heart failure presented at Emergency of a tertiary care hospital
30-day Prognosis | From day of admission of last visit till 30 days
  Factors affecting the 30-day prognosis of patients with acute heart failure either via telephonic contact or re-admission or via OPD.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Fatima, MBBS, FCPS, Principal Investigator — National Institute of Cardiovascular Diseases
Locations (1):
- National Institute of Cardiovascular Diseases, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
The Hospital Medical Record number will be used as the patient identifier.